CLINICAL TRIAL: NCT00962637
Title: A Phase III, Randomized, Double-Blind, Placebo-Controlled, Open-Label, Active-Controlled Study to Evaluate the Safety and Efficacy of Androxal™ Treatment in Men With Secondary Hypogonadism
Brief Title: Study to Evaluate the Safety and Efficacy of Androxal™ Treatment in Men With Secondary Hypogonadism
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Repros Therapeutics Inc. (Industry)
Responsible Party: Andre van As, MD, PhD, Repros Therapeutics, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZA-003
Record Dates: First submitted 2009-08-18; First posted 2009-08-20 (Estimated); Last update posted 2010-02-11 (Estimated); Status verified 2010-02

CONDITIONS: Secondary Hypogonadism
Keywords: Secondary Hypogonadism
MeSH Terms: conditions — Hypogonadism | interventions — Enclomiphene; Testosterone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): Androxal™ 12.5 mg
  Interventions: Drug: Androxal
- 2 (Experimental): Androxal™ 25 mg
  Interventions: Drug: Androxal
- 3 (Active Comparator): AndroGel®
  Interventions: Drug: AndroGel
- 4 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Androxal — 12.5 mg once daily
  Other Names: Enclomiphene citrate
  Arms: 1
Drug: Androxal — 25 mg once daily
  Other Names: Enclomiphene citrate
  Arms: 2
Drug: AndroGel — 5 g applied topically daily. The subject was to return to the clinic every 2 weeks for the first 2 months to monitor serum testosterone levels. If testosterone concentration remained below the normal level, the dose of AndroGel® could have been increased to 10 g and then to 15 g according to the guidance provided in the product package insert.
  Arms: 3
Drug: Placebo — 1 capsule daily
  Arms: 4

SUMMARY:
Approximately 4 to 5 million men in the U.S. are testosterone-deficient. Enclomiphene (trans-clomiphene) citrate (Androxal) was evaluated to determine if Androxal increased serum testosterone levels in men with secondary hypogonadism. Subjects were randomly assigned to 1 of 4 treatments groups. Appropriate amounts of medications were dispensed at each visit. Subjects took their medications orally or by rubbing it onto the skin (depending on the treatment assignment) once daily for up to 6 months. Treatment visits occurred at approximately 4-week intervals for Months 1, 2, and 3 and then at 6-week intervals for Months 4, 5, and 6.

ELIGIBILITY:
Inclusion Criteria:

* Total serum testosterone concentrations < 300 ng/dL at baseline

Exclusion Criteria:

* Presence or history of prostate cancer
* Elevated PSA > 3.5 ng/mL

Additional inclusion and exclusion criteria may apply.

Ages: 18 Years to 68 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2006-03; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety of Androxal™ administered in men with secondary hypogonadism | Six months

SECONDARY OUTCOMES:
Demonstrate that treatment of men with secondary hypogonadism with Androxal™ was non-inferior to treatment with the active control, AndroGel® | Six months

CONTACTS AND LOCATIONS:
Overall Officials: Andre van As, MD, PhD, Study Director — Repros Therapeutics Inc.
Locations (18):
- United States (18):
  - Alabama Clinical Therapeutics, LLC, Birmingham, Alabama
  - Medical Affiliated Research Center, Inc., Huntsville, Alabama
  - Northern California Research Corp., Carmichael, California
  - Prime-Care Clinical Research, Mission Viejo, California
  - Harbor-UCLA Medical Center, Torrance, California
  - Chase Medical Research, LLC, Waterbury, Connecticut
  - Southeastern Research Group, Inc., Tallahassee, Florida
  - Northeast Indiana Research, LLC, Fort Wayne, Indiana
  - Commonwealth Biomedical Research, Madisonville, Kentucky
  - The Center for Sexual Medicine at Sheppard Pratt, Baltimore, Maryland
  - Office of Keith Pierce, MD, Livonia, Michigan
  - Office of Michael Mall, MD, Las Vegas, Nevada
  - Office of Stephen Miller, MD, Las Vegas, Nevada
  - Advanced Biomedical Research, Inc., Hackensack, New Jersey
  - Office of Gary S. Karlin, Lawrenceville, New Jersey
  - Medial Research Associates of Nashville, Nashville, Tennessee
  - Urology San Antonio Research, PA, San Antonio, Texas
  - Salt Lake Research, Salt Lake City, Utah